CLINICAL TRIAL: NCT02822911
Title: Benefit of Carbohydrate Deficient Transferrin to Detect Chronic Alcohol Abuse in the Elderly. A French Multicentered Prospective Interventional Study.
Brief Title: Benefit of Carbohydrate Deficient Transferrin to Detect Chronic Alcohol Abuse in the Elderly
Acronym: Caesar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GHRMSA 809; 2016-A00027-44 (Other: France: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2016-11

CONDITIONS: Alcohol Abuse
Keywords: elderly; chronic alcoholism; Carbohydrate Deficient Transferrin; Biological Detection / Diagnosis
MeSH Terms: conditions — Alcoholism; Disease | interventions — Ethanol; carbohydrate-deficient transferrin; gamma-Glutamyltransferase; Erythrocyte Indices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alcohol Used Disorders Identification Test (AUDIT C) (Other): Submission of Audit-C questionnaire to all the patients of the study. When the result to the AUDIT-C questionnaire reaches at least 1 point, the analysis of the Carbohydrate deficient transferrin (CDT) is performed within 3 days after the beginning of the study. Results of Gamma glutamyl transpeptidase (GGT) and Mean Corpuscular Volume (MCV) performed as routine practice collected at the same time as the CDT analysis.
  Interventions: Behavioral: Alcohol Used Disorders Identification Test (AUDIT C); Procedure: Carbohydrate deficient transferrin; Procedure: Gamma glutamyl transpeptidase; Procedure: Mean Corpuscular Volume

INTERVENTIONS:
Behavioral: Alcohol Used Disorders Identification Test (AUDIT C) — The Audit-C questionnaire is a three item alcohol screen that can help identify persons who are hazardous drinkers or have active alcohol abuse disorders (including alcohol abuse or dependence). The AUDIT-C is a modified version of the 10 question AUDIT instrument.
  Score from 0 to 12. Each Audit-C question has a 5 answer choice, allotted points are from 0 to 4 points. In men, a score of 4 is considered as positive, optimal for identifying hazardous users or active alcohol abuse disorders. The same for 3 points in women.
  Other Names: Audit-C questionnaire
Procedure: Carbohydrate deficient transferrin — Blood sample to collect carbohydrate deficient transferrin (CDT) only if the Alcohol Used Disorders Identification Test (AUDIT C) reports at least 1 point.
  Other Names: CDT
Procedure: Gamma glutamyl transpeptidase — Results of Gamma glutamyl transpeptidase (GGT) performed as routine practice collected only if the Alcohol Used Disorders Identification Test (AUDIT C) reaches at least 1 point.
  Other Names: GGT
Procedure: Mean Corpuscular Volume — Results of Mean Corpuscular Volume (MCV) performed as routine practice collected only if the Alcohol Used Disorders Identification Test (AUDIT C) reports at least 1 point.
  Other Names: MCV

SUMMARY:
Alcohol misuse affects 5 million people in France. Even though the elderly are also concerned by this pathology, there is not much information about chronic alcohol misuse of this population in particular.

Biological markers like gamma-glutamyltranspeptidase (GGT), mean corpuscular volume (MCV) and carbohydrate deficient transferrin (CDT) are usually used to detect alcohol abuse. As a biological marker of alcohol misuse, the specificity of the CDT is known to be superior to the GGT as well.

However, when it comes to the elderly, alcoholism diagnosis tools are based on research of younger populations.

This study aims to evaluate the benefit of the CDT to detect chronic alcohol use in the elderly.

DETAILED DESCRIPTION:
Problematic alcohol misuse is frequent but tends to decrease with age. According to the French Alcohology Society, 10% of the adult population is alcohol abstinent and after 65 years old, they are 40% to abstain from alcohol.

On the other hand, the French Alcohology Society also reports that a regular or daily alcohol consumption for older people increases the risk of dependence on alcohol.

For the elderly, biological disorders can be related to polymedication or other conditions related to the aging process, making it difficult to diagnose alcoholism for aged people.

For the study, the three-item Alcohol Use Disorders Identification Test (AUDIT-C) will be submitted to :

* every patient admitted in the Hospital of Mulhouse (France) for at least a day in the Geriatrics Department
* every patient entering the General Practitioner Support Association of Alsace, France (translated in French as the "RAG").

When the score of the AUDIT-C reaches at least 1 point, the study will collect results of the GGT and MCV performed as routine practice and add the CDT in the blood tests.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years old
* Patients hospitalized for a day or more in the Geriatrics Department of Mulhouse, GHRMSA :

  * Coming from home within 48 hours after admission to the GHRMSA
  * Study procedures performed within 72 hours after admission to the GHRMSA
* Or new members of the General Practitioner Support Association of Alsace, France (translated in French as the "RAG") living in Mulhouse, Thann and Saint Louis cities (France) :

  * Living at home and joining the RAG between the 1st of March and the 31st of October 2016
  * Study Procedures performed within 3 days after enrollment in the study
* Relative or helper available who usually visits the patient at home at least once a week
* Absence of alcoholic excipient in the concomitant medication

Exclusion Criteria:

* Age < 60 years old
* Admitted in the Geriatrics Department of Mulhouse after more than 48hours after admission to the GHRMSA
* Presence of the following symptoms :

  * Hepatobiliary deficiency related to a primary biliary cirrhosis
  * Autoimmune or viral cirrhosis
  * Hepatocellular carcinoma
  * Congenital metabolic disorder in protein glycosylation
* Known genetics variance in Tf B or D transferrin
* Living in an elderly care institution
* Already enrolled in this study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Benefit of Carbohydrate Deficient Transferrin to detect chronic alcohol abuse in the elderly compared to usual clinical detection tools | Within 3 days after enrollment in the study
  Analysis performed when at least 1 point at the AUDIT-C questionnaire, confirming presence of alcohol consumption

SECONDARY OUTCOMES:
Sensitivity and specificity of the disturbance of Gamma-glutamyltranspeptidase when presence of alcohol consumption, with at least 1 point in the AUDIT-C questionnaire | Within 3 days after enrollment in the study
  If collected as routine practice : at the same time as Carbohydrate Deficient Transferrin analysis when Audit-C questionnaire reports at least 1 point
Sensitivity and specificity of the disturbance of Mean Corpuscular Volume when presence of alcohol consumption, with at least 1 point in the AUDIT-C questionnaire | Within 3 days after enrollment in the study
  If collected as routine practice : at the same time as Carbohydrate Deficient Transferrin analysis when Audit-C questionnaire reports at least 1 point
Socio-economic characteristics of alcohol abusers : Socioprofessional category | Within 3 days after enrollment in the study
  Classification of professions and socioprofessional categories of the French National institute of Statistics and economics. 9 types of working classes.
Socio-economic characteristics of alcohol abusers : Education Category | Within 3 days after enrollment in the study
  6 levels of education type, from no degree or 9th grade, to Doctor of Philosophy (PhD). Classification created by the French National institute of Statistics and economics
Socio-economic characteristics of alcohol abusers : Way of life | Within 3 days after enrollment in the study
  Description of the patient's environment :
  * married or not
  * living alone or not
  * professional help provided at home by either a nurse, or cleaning lady, or meal delivery, or senior helper

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Schnell, MD, Principal Investigator — Groupe Hospitalier de la Region de Mulhouse et Sud Alsace
Locations (2):
- France (2):
  - Reseau d'Appui aux Generalistes (RAG), Colmar
  - GHRMSA, Mulhouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnell C (2016) Benefit of carbohydrate deficient transferrin in detecting chronic alcohol abuse in the elderly: study protocol for a multicentre, non-randomized, open-label study. Clin Transl Degener Dis 1(3):121-126.
- See also: Study Protocol — https://www.researchgate.net/publication/308755873_Benefit_of_carbohydrate_deficient_transferrin_in_detecting_chronic_alcohol_abuse_in_the_elderly_study_protocol_for_a_multicentre_non-randomized_open-label_study